CLINICAL TRIAL: NCT06713681
Title: Trop2-targeting the Second Near Infrared (NIR-II) Molecular Probe for the in Vitro Evaluation of Breast Cancer Surgical Margin and Sentinel Lymph Node Metastasis Status
Brief Title: Trop2-targeting NIR-II Molecular Probe for Breast Cancer Precise Surgery
Acronym: NIR-II
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2024-140
Record Dates: First submitted 2024-07-21; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Margins of Excision
Keywords: NIR-II; Trop2; Surgical navigation; Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TTP-ICG incubation: The fresh excision breast masses or lymph nodes will be completely soaked in the TTP-ICG incubation solution (5, 10, 20 μg/mL) for 3, 5, or 10 min, followed by 5 min of rinsing with PBST buffer and drying with absorbent paper.The NIR-II fluorescence imaging will be then performed under the DPM NIR-II system. And the correlation between pathological characterization and fluorescent information will be further analyzed.
  Interventions: Diagnostic Test: TTP-ICG incubation solution

INTERVENTIONS:
Diagnostic Test: TTP-ICG incubation solution — Fresh breast massed and lymph nodes will be incubated with TTP-ICG with different concentrations and times

SUMMARY:
Positive surgical margins are closely associated with local recurrence in breast-conserving surgery (BCS). Meanwhile, accurately assessing sentinel lymph node (SLN) metastasis is crucial for determining the extent of axillary lymph node dissection (ALND) and minimizing complications. Indocyanine green (ICG)-based the second near-infrared (NIR-II) fluorescence imaging offers real-time visualization during surgery, potentially reducing positive margin rates and improving SLN detection, while the specificity remains a challenge. Herein, the investigators will introduce a novel NIR-II probe, TTP-ICG, based on a Trop2-targeting peptide and an approach which enables rapid differentiation between cancer and para-cancer tissue as well as metastatic and normal lymph nodes. In brief, fresh tissues will be soaked in TTP-ICG immediately after resection, and their histological characterization will be determined under NIR-II fluorescence imaging. Pathological confirmation will further validate our approach.

DETAILED DESCRIPTION:
After patient enrollment, surgical treatment will be administered based on clinical diagnosis and treatment. During the surgery, excised breast masses or lymph nodes will undergo incubation with TTP-ICG following this specific procedure:

1. Preparation of the incubation solution: TTP-ICG will be dissolved in phosphate-buffered saline (PBS) at room temperature in the dark, with varying concentrations (5, 10, 20 μg/mL).
2. Incubation of fresh breast masses or lymph nodes: The freshly excised breast masses or lymph nodes will be immersed and gently agitated in the incubation solution for 3, 5, or 10 minutes. Subsequently, they will be rinsed with PBST buffer (PBS with Tween 20) for 5 minutes and dried using absorbent paper.
3. Acquisition of NIR-II images: NIR-II images and fluorescent intensities will be captured using the "Digital Precision Medicine (DPM)" NIR-II system, optimized with appropriate parameters.
4. Pathological diagnosis and data analysis: Hematoxylin and eosin staining, along with immuno-histochemistry, will be performed. The subsequent correlation between pathological characterization and fluorescent information will be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-75 years of age
* Female
* Patients presenting with a breast nodule or mass presumed to be resectable on pre-operative assessment
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Patients unable to participate in the consent process
* Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc
* Other conditions that the researcher considers inappropriate to participate in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 40 female patients, aged 18 to 75 years, who have been assessed to have resectable breast nodules or masses and are scheduled to undergo surgery. During the surgery, the resected tumors and lymph nodes will be incubated with the TTP-ICG solution, and NIR-II fluorescence signals from the tissues will be collected.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differentiation of breast cancer, para-cancer tissues, and benign masses as well as metastatic and normal lymph nodes | 1 year
  NIR-II fluorescence intensity of breast cancer, para-cancer tissues, and benign masses as well as metastatic and normal lymph nodes after TTP-ICG incubation .
Expression of the Trop-2 in the breast cancer and metastatic lymph nodes | 1 year
  NIR-II fluorescence intensity of the breast cancer tissues and metastatic lymph nodes with different Trop-2 expression level after TTP-ICG incubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Zhang Y, Zhang L, Luo X, Yang X, Zhu Y, Wang G, Huang W, Zhang D, Zeng Y, Li R, Guo C, Wang J, Wu Z, Liu N, Zhang G. Intraoperative evaluation of tumor margins using a TROP2 near-infrared imaging probe to enable human breast-conserving surgery. Sci Transl Med. 2024 Oct 16;16(769):eado2461. doi: 10.1126/scitranslmed.ado2461. Epub 2024 Oct 16. PMID 39413161